CLINICAL TRIAL: NCT05134545
Title: A Multicenter, Prospective, Randomized, Double-blind, Pivotal Clinical Study to Evaluate the Effectiveness and Safety of GENOSS® DCB Versus IN.PACT Admiral® DCB in Patients With Peripheral Artery Disease of Femoral and Popliteal Artery
Brief Title: Compare the Effectiveness and Safety of Genoss® DCB and IN.PACT Admiral® DCB in Patients With Peripheral Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genoss Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSP-DS1411
Record Dates: First submitted 2021-11-02; First posted 2021-11-26 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Peripheral Artery Disease; De Novo Stenosis
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genoss® DCB (Experimental): Paclitaxel Coated PTA Balloon Catheter
  Interventions: Device: Genoss® DCB
- IN.PACT Admiral® DCB (Active Comparator): Paclitaxel Coated PTA Balloon Catheter
  Interventions: Device: IN.PACT Admiral® DCB

INTERVENTIONS:
Device: Genoss® DCB — Peripheral Drug Coated Balloon
  Arms: Genoss® DCB
Device: IN.PACT Admiral® DCB — Peripheral Drug Coated Balloon
  Arms: IN.PACT Admiral® DCB

SUMMARY:
The purpose of this clinical trial is to demonstrate the non-inferiority of GENOSS DCB versus IN.PACT Admiral DCB on late lumen loss 6 months after the procedure in patients with de novo or non-stented restenotic lesions of the superficial femoral artery and popliteal artery and to evaluate the safety.

This clinical trial will be conducted on a total of 118 patients at 11 domestic institutions (taking into account the dropout rate of 30%).

DETAILED DESCRIPTION:
In this clinical trial, IN.PACT Admiral, which is the most similar to GENOSS DCB, a test device, and the product type and purpose of use, and whose effectiveness has already been proven through numerous clinical studies, was selected as a control product.

Due to the nature of this clinical trial, the investigator cannot be blinded to the treatment method to which the subject is assigned, so it is designed as a double-blind design in which only the subject and the independent evaluator are blinded.

For efficacy and safety evaluation, follow-up is performed up to 12 months after procedure of the clinical trial medical device.

The primary endpoint of the effectiveness evaluation was performed by an independent evaluator and CT angiography at 6 months of in-segment late lumen loss.

It is evaluated the revascularization rate, Rutherford classification, the amount of change in ABI or TBI at 1, 6, and 12 months, the procedural success rate during the clinical trial period, and the device success rate immediately after the procedure.

Safety evaluation is confirmed through all adverse events, MAE (Major adverse event), vital signs, physical examination and laboratory test results that occur to the subject during the clinical trial period after procedure of the clinical trial medical device.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 19 years and ≤ 85 years of age
2. Documented ischemia with Rutherford classification 2, 3, 4 or 5
3. Target lesion is in the SFA and/or PPA
4. Reference vessel diameter ≥ 4 mm and ≤ 7 mm by visual estimate
5. Angiographic evidence that target lesion consists of a single de novo or non-stented restenotic lesion;

   * 70% - 99% occluded with total lesion length ≥ 40 mm and ≤ 300 mm
   * 100% occluded with total lesion length ≤ 100 mm
   * Combination lesions (a non-occlusive lesion that includes a totally occluded segment along its length) are eligible provided that (1) the combined lesion length is ≥ 40 mm and ≤ 300 mm and (2) the totally occluded segment is not greater than 100 mm in length.
   * Tandem or adjacent lesions are treated as a single lesion, the gap between the lesions is ≤ 30 mm, and the total combined lesion length including the distance between the lesions is ≥ 40 mm and ≤ 300 mm

Exclusion Criteria:

1. Stroke or STEMI within 3 months prior to enrollment
2. Acute thrombosis or acute aneurysm in the target lesion
3. History of or planning to have a major amputation in the leg
4. Failure to successfully cross the target lesion with a guidewire
5. Poor distal run-off artery to the ankle or lower
6. Known allergies or sensitivities to paclitaxel, shellac, vitamin E, heparin, aspirin, other anticoagulant/antiplatelet therapies or contrast agent
7. Target lesion is one of the following;

   * In-stent restenosis (ISR)
   * Restenosis after DCB procedure
   * Previously treated with bypass surgery
   * Severe concentric calcified lesions on angiography where pre-dilation cannot be performed or failed, and the procedure for the device for clinical trials is inadequate
8. Those who need stenting due to vascular dissection that restricts blood flow of Grade D or higher after pre-dilation
9. Any major (e.g., cardiac, peripheral, abdominal) intervention (including in the contralateral SFA/PPA) planned within 30 days post index procedure
10. Life expectancy, in the Investigator's opinion, is less than 12 months
11. Chronic renal insufficiency with serum creatinine > 2.5 mg/dL

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2019-03-24 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
late lumen loss after procedure in patients with peripheral artery disease of femoral and popliteal artery | Follow-up CT angiography at 6 months after the procedure
  late lumen loss between test group and control group evaluated by CT angiography in patients with peripheral artery disease of femoral and popliteal artery

SECONDARY OUTCOMES:
Target lesion revascularization | at 1 months, 6 months, and 12 months after procedure
  Proportion of subjects who underwent revascularization because the ABI (or TBI) decreased by 20% or more, or exceeded 0.15, or showed clinically significant ischemic symptoms compared to immediately after the procedure
Change in ABI or TBI | at 1 month, 6 months, and 12 months after procedure
  The amount of ABI(Ankle-brachial index) or TBI(Toe-brachial index) change after the procedure compared to before the procedure is evaluated between the test group and the control group.
Changes in Rutherford classification | at 1 month, 6 months, and 12 months after procedure
  The amount of change in Rutherford classification after the procedure compared to before the procedure is evaluated between the test group and the control group.
Restenosis rate after procedure in patients with peripheral artery disease of femoral and popliteal artery | Follow-up CT angiography at 6 months after procedure
  Restenosis is defined as a case where the DS(Diameter stenosis) of the reference vessel diameter is 50% or more when the successfully treated lesion is evaluated through CT angiography.
Device success rate, % | immediately after the procedure
  It is defined as a device that has successfully reached the target lesion during the procedure, undergoes normal balloon inflation and deflation, and is fully recovered without balloon rupture.
Procedural success rate, % | at 12 months after procedure
  During the clinical trial period, no postoperative death, target vessel revascularization (TVR), lower extremity amputation, or target lesion thrombosis is defined as procedural success.

CONTACTS AND LOCATIONS:
Overall Officials: Je Hwan Won, MD, Principal Investigator — Department of Radiology, Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, South Korea